CLINICAL TRIAL: NCT06006871
Title: The Secret Trail of Moon (MOON): a Personalized Treatment Video Game for Children and Adolescents With ADHD Based on Cognitive Training and Self-regulation
Brief Title: Effectiveness of the Serious Video Game MOON in Emotional Regulation in ADHD
Acronym: MOON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Hilario Manuel Blasco Fontecilla, Child and adolescent psychiatrist, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI 106/22; IND2020/BMD-17544 (Other Grant/Funding Number: Community of Madrid); Expte. 1061/22/EC-R. (Other: Spanish Agency of Medicines and Medical Devices (AEMPS))
Record Dates: First submitted 2023-05-07; First posted 2023-08-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized, unblinded, PRE-POST intervention study with concealment of the randomization sequence.
  A randomization of 2 groups by blocks will be performed: Group 1: "The Secret Trail of Moon" (MOON): a personalized cognitive training with a face-to-face and online video game (n=76); Group 2: Passive control (TAU): usual treatment (pharmacological) without cognitive training intervention (n=76).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Secret Trail of Moon (MOON): Cognitive training with Serious Video Game (Experimental): The Secret Trail of Moon is a therapeutic video game that has been created for the cognitive training of patients with ADHD. Five mechanisms have been designed to work on five cognitive functions that are deficient in ADHD: sustained attention, working memory, reasoning, planning and visuospatial ability. Aspects of rewards and music therapy have been added to this enhanced version of the game.
  In this second clinical trial, the impact has been extended to twice a week during 20 sessions. There are two platforms of the same version of the game: computer (7-11 years old) and virtual reality (12-18 years old). Patients have to come to the hospital twice a week for training sessions of about 20-30 minutes duration for 10 weeks. Subsequently, they are given the computer version of the video game on a USB so that they can play it at home for another 10 weeks (twice a week).
  Participants are monitored for possible difficulties and/or side effects.
  Interventions: Behavioral: The Secret Trail of Moon (MOON): Cognitive training with Serious Video Game; Drug: Usual treatment for ADHD
- Control Group (Active Comparator): This group corresponds to the control group (n=76). The control group continues with their prescribed pharmacological treatment without any cognitive intervention.
  The participants of this group are contacted by telephone once a week to follow up on possible difficulties and/or side effects.
  Interventions: Drug: Usual treatment for ADHD

INTERVENTIONS:
Behavioral: The Secret Trail of Moon (MOON): Cognitive training with Serious Video Game — Patients are pharmacologically stable and receive a cognitive intervention with our videogame twice a week in the hospital (10 sessions) and twice a week in their home with a computer video game (other 10 sessions).
  Arms: The Secret Trail of Moon (MOON): Cognitive training with Serious Video Game
Drug: Usual treatment for ADHD — All patients continue with their stable pharmacological treatment and do not receive any additional cognitive intervention.

SUMMARY:
Introduction: Attention Deficit Hyperactivity Disorder (ADHD) is the most common neurodevelopmental disorder in childhood and adolescence (5%) with associated difficulties and worse prognosis if undetected. Multimodal treatment is the treatment of choice, however, sometimes it can be insufficient or have some drawbacks.

Objective: To demonstrate the effectiveness of cognitive training through the video game 'The Secret Trail of Moon' (MOON) in improving emotional regulation of ADHD in people aged 7 to 18 years.

Hypotheses: H1: ADHD patients using MOON improve their emotional regulation more than the control group; H2: ADHD patients using MOON improve in symptomatology with respect to the control group; H3: ADHD patients using MOON improve their cognitive abilities than the control group; H4: ADHD patients using MOON improve in academic performance with respect to the control group; H5: The change of platform (face-to-face, online) does not entail differences in emotional regulation; H6: There are no side effects associated with the video game.

Methods: Design: prospective, unicenter, randomized, unblinded, PRE-POST intervention study. Randomization of the groups (MOON vs. Control) will be performed by electronic CRD. The MOON intervention will be performed 2 times/week for 10 weeks (30 minutes/session). The first five weeks (10 sessions) will be conducted face-to-face; the remaining weeks will be conducted online at the participants' home.

Sample: 152 patients with a clinical diagnosis of ADHD (CGI between 3 and 6) with pharmacological treatment.

Evaluation: a data collection notebook will be used to obtain demographic and clinical data. The data will be recorded with electronic CRD (REDCap). Measures to answer the hypotheses will be made through clinical scales for parents and objective tests of cognitive abilities in patients. Additional information on academic performance will be collected.

Statistical power analysis: The study has a power greater than 80% to detect differences.

Statistical analysis: Classical statistics: T student, 2-factor ANOVA and Mann Whitney analyses will be performed according to the characteristics of each variable.

Ethics: The study was approved by the Research Ethics Committee of the Hospital Universitario Puerta de Hierro on December 14th, 2022. The authorization of the Spanish Agency of Medicines and Health Products was February 14th, 2023. Informed consent will be requested from legal guardians and minors protecting their personal data to the provisions of the Organic Law 3/2018 of 5 December, on Personal Data Protection and guarantee of digital rights.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17 years (could turn 18 during the study)
* Clinical diagnosis of ADHD in any presentation.
* With pharmacological treatment for ADHD.
* Ability to follow verbal instructions
* Ability to play a video game (not necessary to play regularly).
* Clinically stable. ADHD symptomatology severity based on clinician-assessed CGI score (between 3-6).

Exclusion Criteria:

* Severe patients (> or equal to 5 CGI) or very mild patients (CGI < or equal to 1)
* Patient at risk of suicide (according to the clinical judgment of the professional in charge of the patient)
* Motor difficulties that prevent playing the videogame
* Participation in other similar studies
* Intention to initiate any psychotherapeutic treatment (including cognitive-behavioral therapy) in the next 3 months of the course of participation in the clinical trial.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Strenghts and difficulties questionnaire (SDQ) for parents | 3 months
  This questionnaire has 25 items (duration of approximately 5 minutes). It mainly measures the scales 1) Emotional symptoms, 2) Behavioral problems, 3) Hyperactivity, 4) Problems with peers and 5) Prosocial behavior. A decrease of 3 to 4 points in the post-assessment visit (D70) with respect to the pre-assessment visit (D0) will be considered an improvement in emotional regulation (Goodman, 1977)

SECONDARY OUTCOMES:
The Swanson, Nolan, and Pelham Rating Scale (SNAP-IV) for parents | 3 months
  The main ADHD symptomatology (inattention, hyperactivity, impulsivity) will be measured with subjective scales for parents. The SNAP IV is a scale for the assessment of ADHD symptoms. It's an 18-item questionnaire with a Likert scale of 0-4 (approximately 5 minutes long) of which 9 assess attention deficit and another 9 assess hyperactive-impulsive component. The cut-off points for attention deficit are 1.78 for parents. For hyperactivity-impulsivity they are 1.44 for parents.
The Conners Abbreviated Symptom Questionnaire (CPRS-HI) for parents | 3 months
  The main ADHD symptomatology (inattention, hyperactivity, impulsivity) will be measured with subjective scales for parents. The Conners scales are a set of scales for the assessment of patients with ADHD. CPRS-HI is a 10-item questionnaire with a Likert scale of 0-3 (approximately 2 minutes long). This revised and abbreviated version of the Conners scale is designed to be answered by parents of children ages 6-18. It consists of 10 items with a Likert type response: 0= not true at all/never; 1= just a little true/occasionally; 2= Pretty much true/often; 3=very much true/very often.
  The cut-off points are divided by gender. For children, a score above 16 is suspected ADHD. While for girls, a suspected diagnosis of ADHD is from 12 points
Clinical Global Impression Scale (CGI) for parents | 3 months
  Symptom severity will be measured with the Clinical Global Impression Scale (CGI) adaptation for parents of approximately 1 minute duration, consisting of a "thermometer" with a Likert scale of 1-10.
The Sleep Disturbance Scale for Children (SDSC) for parents | 3 months
  Sleep difficulties will be measured with the Sleep Disturbance Scale for Children (SDSC). It is a 26-item questionnaire with a Likert scale of 1-5 (1: never; 5: always) with an approximate duration of 5 minutes (Bruni et al., 1996)
Behavior Rating Inventory Executive Function 2 (BRIEF-2) questionnaire for parents | 3 months
  Executive dysfunction will be evaluated by means of subjective scales for parents and objective tests for patients. The subjective test for parents will be performed with the Behavior Rating Inventory Executive Function 2 (BRIEF-2) questionnaire.The BRIEF-2 is a questionnaire designed for the evaluation of executive functions in children and adolescents. It is made up of 63 items with three answer options (never, sometimes and frequently). Its correction provides four general indexes: emotional regulation, cognitive regulation, behavioral regulation and global index of executive function.
Conners Continuous Performance Test 3rd Edition (CPT-3) for patients with ADHD | 3 months
  Executive dysfunction will be evaluated by means of subjective scales for parents and objective tests for patients. Conners Continuous Performance Test-3 (CPT-3) is a task that is usually used to screen for ADHD in addition to measuring sustained attention, impulse control and processing speed. The Conners CPT-3 is a computerized, standardized, and validated application test for different age and gender groups. The test consists of pressing a button each time a letter (target) appears on the screen, except for the letter X (non-target), which should not be pressed. The duration is approximately 14 minutes and the presentation interval between letters is variable (1, 2 and 4 seconds). The test provides results on hits, error of omission (undetected target) and errors of commission (reacted non-target), which are considered a measure of impulsivity. In addition, CPT3-3 provides information on mean reaction time and reaction time variability of hits.
Corsi Cubes for patients with ADHD | 3 months
  Executive dysfunction will be evaluated by means of subjective scales for parents and objective tests for patients. Corsi Cubes to measure visuospatial working memory (Corsi, 1972; Kessels et al., 2000)
Comprehensive Trail-Making Test Second Edition (CTMT-2) for patients with ADHD | 3 months
  Executive dysfunction will be evaluated by means of subjective scales for parents and objective tests for patients. Comprehensive Trail-Making Test Second Edition (CTMT-2) to measure cognitive flexibility, with three indexes: inhibitory control, task switching and total index.
Game Addiction Scale for Adolescents (GASA) for patients with ADHD | 3 months
  Game Addiction Scale for Adolescents (GASA) is a 7-item questionnaire to assess video game addiction (Lemmens et al., 2009)
Academic notes | 3 months
  Information about academic performance will be obtained with grades.
"Clinical Examinations Questionnaire"(UKU) for patients with ADHD | 3 months
  UKU is a tool designed to evaluate possible secondary symptoms that happen during the week. This scale is not included in the assessment phases. Only the MOON with VR group should complete the scale after each cognitive training session.

OTHER OUTCOMES:
Clinical Global Impression Scale (CGI) for clinicians | 3 months
  Symptom severity will be measured with the Clinical Global Impression Scale (CGI) approximately 1 minute duration. ADHD symptomatology severity based on clinician-assessed CGI score (between 3-6) for inclusion criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Puerta de Hierro University Hospital, Majadahonda, Madrid, Spain

REFERENCES:
- [Background] Rodrigo-Yanguas M, Martin-Moratinos M, Menendez-Garcia A, Gonzalez-Tardon C, Sanchez-Sanchez F, Royuela A, Blasco-Fontecilla H. A Virtual Reality Serious Videogame Versus Online Chess Augmentation in Patients with Attention Deficit Hyperactivity Disorder: A Randomized Clinical Trial. Games Health J. 2021 Aug;10(4):283-292. doi: 10.1089/g4h.2021.0073. PMID 34370610
- [Result] Rodrigo-Yanguas M, Martin-Moratinos M, Menendez-Garcia A, Gonzalez-Tardon C, Royuela A, Blasco-Fontecilla H. A Virtual Reality Game (The Secret Trail of Moon) for Treating Attention-Deficit/Hyperactivity Disorder: Development and Usability Study. JMIR Serious Games. 2021 Sep 1;9(3):e26824. doi: 10.2196/26824. PMID 34468332
- [Result] Rodrigo-Yanguas M, Martin-Moratinos M, Gonzalez-Tardon C, Sanchez-Sanchez F, Royuela A, Bella-Fernandez M, Blasco-Fontecilla H. Effectiveness of a Personalized, Chess-Based Training Serious Video Game in the Treatment of Adolescents and Young Adults With Attention-Deficit/Hyperactivity Disorder: Randomized Controlled Trial. JMIR Serious Games. 2023 Apr 24;11:e39874. doi: 10.2196/39874. PMID 37093628
- [Result] Sujar A, Martin-Moratinos M, Rodrigo-Yanguas M, Bella-Fernandez M, Gonzalez-Tardon C, Delgado-Gomez D, Blasco-Fontecilla H. Developing Serious Video Games to Treat Attention Deficit Hyperactivity Disorder: Tutorial Guide. JMIR Serious Games. 2022 Aug 1;10(3):e33884. doi: 10.2196/33884. PMID 35916694
- [Result] Bella-Fernandez M, Martin-Moratinos M, Li C, Wang P, Blasco-Fontecilla H. Differences in Ex-Gaussian Parameters from Response Time Distributions Between Individuals with and Without Attention Deficit/Hyperactivity Disorder: A Meta-analysis. Neuropsychol Rev. 2024 Mar;34(1):320-337. doi: 10.1007/s11065-023-09587-2. Epub 2023 Mar 6. PMID 36877328
- [Derived] Martin-Moratinos M, Bella-Fernandez M, Rodrigo-Yanguas M, Gonzalez-Tardon C, Li C, Wang P, Royuela A, Lopez-Garcia P, Blasco-Fontecilla H. Effectiveness of a Virtual Reality Serious Video Game (The Secret Trail of Moon) for Emotional Regulation in Children With Attention-Deficit/Hyperactivity Disorder: Randomized Clinical Trial. JMIR Serious Games. 2025 Jan 8;13:e59124. doi: 10.2196/59124. PMID 39773848
- [Derived] Martin-Moratinos M, Bella-Fernandez M, Rodrigo-Yanguas M, Gonzalez-Tardon C, Sujar A, Li C, Wang P, Royuela A, Lopez-Garcia P, Blasco-Fontecilla H. Effectiveness of a Serious Video Game (MOON) for Attention Deficit Hyperactivity Disorder: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2024 Feb 23;13:e53191. doi: 10.2196/53191. PMID 38393773